CLINICAL TRIAL: NCT07243951
Title: Phase II Clinical Study on the Efficacy and Safety of the Combination of Cadonilimab and Capecitabine in Adjuvant Therapy for Combined Hepatocellular Carcinoma and Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-381R
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Combined Hepatocellular-cholangiocarcinoma; Liver Neoplasms
Keywords: Cadonilimab; Capecitabine; Phase II Clinical Trial; Bispecific Antibody; PD-1; CTLA-4; Recurrence-Free Survival; Immunotherapy; Adjuvant Therapy
MeSH Terms: conditions — Liver Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab + Capecitabine Combination Therapy (Experimental): This arm receives the combination therapy of Cadonilimab (intravenous infusion, 10 mg/kg, once every 3 weeks) and Capecitabine (oral, 2500 mg/m²/day administered in two divided doses, on a schedule of 2 weeks of treatment followed by 1 week of rest) for up to 8 cycles (24 weeks), or until disease recurrence, unacceptable toxicity, or other treatment discontinuation criteria are met.
  Interventions: Drug: Cadonilimab; Drug: Capecitabine

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab is a bispecific monoclonal antibody targeting both PD-1 and CTLA-4. It will be administered intravenously at a dose of 10 mg/kg over 60-120 minutes (no less than 60 minutes) on Day 1 of each 3-week cycle.
Drug: Capecitabine — Capecitabine is an oral chemotherapeutic prodrug that is converted to 5-fluorouracil in the body. The dose is 2500 mg/m² per day, administered orally in two divided doses (morning and evening) within 30 minutes after a meal. It is given for 2 weeks followed by a 1-week rest, constituting one 3-week cycle.

SUMMARY:
Title: A Study of Cadonilimab Combined with Capecitabine After Surgery for Mixed Type Liver Cancer

This is a phase II clinical trial. The main purpose of this study is to find out if using two drugs together, cadonilimab (an immunotherapy drug) and capecitabine (a chemotherapy drug), can help prevent the cancer from coming back after surgery in patients with a specific type of liver cancer called combined hepatocellular-cholangiocarcinoma (cHCC/CCA). This type of liver cancer is rare and has a high chance of returning even after successful surgery.

The study will involve about 75 patients who have had their tumor completely removed but are still at medium to high risk of the cancer returning. All participants in the study will receive the same combination of drugs. Cadonilimab is given through a vein every three weeks. Capecitabine is taken as a pill twice a day for two weeks, followed by one week off. This cycle repeats for up to 8 cycles (about 6 months), or until the cancer comes back or side effects become too severe.

Researchers will primarily measure how long patients live without the cancer returning (Recurrence-Free Survival). They will also track how long patients live overall (Overall Survival), and carefully record any side effects to understand the safety of this treatment combination.

The study hypothesis is that this combination therapy will significantly prolong RFS compared to historical outcomes with surgery alone, while demonstrating acceptable safety.

DETAILED DESCRIPTION:
Protocol Title: Phase II Clinical Trial on the Efficacy and Safety of the Combination of Cadonilimab and Capecitabine in Adjuvant Therapy for Combined Hepatocellular Carcinoma and Intrahepatic Cholangiocarcinoma

Study Background and Rationale:

Combined hepatocellular-cholangiocarcinoma (cHCC/CCA) represents a rare primary liver malignancy exhibiting dual hepatocellular and cholangiocellular differentiation, accounting for approximately 0.4%-14.2% of all liver cancers. Despite R0 resection, postoperative recurrence rates remain exceedingly high (78.6% in reported series), with median overall survival of only 9-18 months. Currently, no standardized adjuvant therapy exists for cHCC/CCA following resection. This study investigates a novel combination strategy utilizing cadonilimab (a bispecific antibody targeting both PD-1 and CTLA-4) with capecitabine chemotherapy to address this unmet medical need by potentially enhancing antitumor immunity and eliminating micrometastatic disease in the postoperative setting.

Study Design:

This is a prospective, single-arm, open-label, multi-center phase II clinical study conducted under investigator initiation.

Intervention Protocol:

* Cadonilimab (AK104): 10 mg/kg administered via intravenous infusion over 60-120 minutes (minimum 60 minutes) on Day 1 of each 21-day cycle.
* Capecitabine: 2500 mg/m²/day administered orally in two divided doses within 30 minutes after morning and evening meals for 14 consecutive days followed by 7 days rest, constituting one 21-day cycle.
* Treatment Duration: Treatment continues for 8 cycles (24 weeks) unless terminated earlier due to: radiologically confirmed disease recurrence per RECIST 1.1, unacceptable toxicity, withdrawal of consent, or investigator decision.

Study Assessments:

* Tumor Evaluations: Radiological assessments (CT/MRI) performed every 12 weeks (4 cycles) during treatment. Post-treatment, patients without recurrence undergo imaging every 12 weeks until 24 months, followed by ultrasonography every 3 months with additional MRI/CT as clinically indicated.
* Safety Monitoring: Comprehensive safety assessments including adverse event monitoring (NCI-CTCAE v5.0), laboratory evaluations (hematology, biochemistry, coagulation, thyroid function), vital signs, physical examinations, and ECG performed at each cycle.
* Follow-up Schedule: Safety follow-up continues for 90 days after last cadonilimab dose or 30 days after last capecitabine dose. Survival follow-up conducted every 3 months (±14 days) via telephone or clinic visit after treatment completion.

Statistical Considerations:

The sample size of 75 patients was calculated to detect an improvement in median RFS from 12.2 months (historical control) to 18 months (HR=0.678) with 80% power at two-sided alpha=0.05, accounting for 5% drop-out rate. Efficacy analyses will utilize the Full Analysis Set (FAS) with Kaplan-Meier methodology for estimating RFS and OS, supplemented with 95% confidence intervals using Clopper-Pearson method.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. ECOG Performance Status ≤ 1.
3. Pathologically confirmed combined hepatocellular carcinoma and intrahepatic cholangiocarcinoma (cHCC/CCA), with R0 resection and classified as Stage IB, Stage II, Stage IIIA, Stage IIIB, or Stage IA (G3) according to AJCC TNM Staging System (8th Edition, 2017).
4. No extrahepatic metastasis.
5. Post-operative Child-Pugh liver function class A; ECOG PS score: 0-1.
6. For subjects with chronic HBV infection, HBV-DNA must be <500 IU/mL. HBsAg-positive patients must receive antiviral therapy according to the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015)". HCV-RNA positive patients must receive antiviral therapy according to the "Guidelines for the Prevention and Treatment of Hepatitis C (2015)" and have normal liver function.
7. Adequate organ function, defined as follows:

(1) Hematological tests (no blood transfusion or use of hematopoietic growth factors within 14 days prior to screening):

1. Hemoglobin (HB) ≥90 g/L
2. Absolute neutrophil count (ANC) ≥1.5×10⁹/L
3. Platelet count (PLT) ≥75×10⁹/L (2) Biochemical tests (no blood transfusion or blood products within 14 days prior to screening):

1) Albumin (ALB) ≥29 g/L 2) ALT and AST <2.5 × ULN 3) Total bilirubin (TBIL) ≤1.5 × ULN 4) Creatinine (Cr) ≤1.5 × ULN (3) International Normalized Ratio (INR) ≤2.3, or Prothrombin Time (PT) prolongation ≤6 seconds beyond the normal control range.

8. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 14 days before initiating study treatment and be willing to use effective and reliable methods of contraception during the trial and for one year after the last dose of the study drug.

9. Subjects voluntarily join the study, sign the informed consent form, have good compliance, and are willing to cooperate with follow-up.

10. No evidence of tumor recurrence or metastasis at baseline examination.

Exclusion Criteria:

1. Pathological diagnosis of hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (ICC), or hilar cholangiocarcinoma.
2. Incomplete tumor resection (non-R0), or postoperative pathology indicating a diagnosis other than cHCC/CCA.
3. History of or concurrent other malignancies, except for cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc. Concurrent autoimmune diseases (e.g., autoimmune liver disease, systemic lupus erythematosus).
4. Child-Pugh class B or C; history or presence of manifestations of hepatic decompensation (e.g., ascites, hepatic encephalopathy, upper gastrointestinal bleeding, etc.).
5. Known hereditary or acquired bleeding or thrombotic tendencies, such as hemophilia.
6. Presence of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 2 months prior to study participation.
7. Myocardial ischemia of grade II or above, myocardial infarction, or poorly controlled arrhythmias (including QTcF interval ≥450 ms for males or ≥470 ms for females; QTc interval calculated by Fridericia's formula). Cardiac insufficiency of NYHA Class III-IV or left ventricular ejection fraction (LVEF) <50% on echocardiography.
8. Severe cardiopulmonary dysfunction or severe renal insufficiency.
9. History of thrombotic/embolic events within the past 6 months, such as cerebrovascular events (including transient ischemic attack) or pulmonary embolism.
10. Inability to swallow, chronic diarrhea, or intestinal obstruction that significantly affects drug administration and absorption.
11. Untreated active hepatitis (Hepatitis B: HBsAg positive with abnormal liver function and HBV-DNA ≥500 IU/mL; Hepatitis C: HCV-RNA positive with abnormal liver function).
12. Human Immunodeficiency Virus (HIV) infection.
13. Active infection or unexplained fever (>38.5°C) occurring during the screening period or before the first dose.
14. Receipt of any vaccine within 30 days prior to enrollment. Planned or prior history of allogeneic organ or bone marrow transplantation, including liver transplantation.
15. History or current presence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function, or other conditions that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
16. Hypertension that cannot be well controlled with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
17. Coagulation dysfunction (PT >16s, APTT >43s, TT >21s, Fibrinogen <2 g/L), bleeding tendency, or ongoing thrombolytic or anticoagulant therapy.
18. Significant clinically significant bleeding symptoms or definite bleeding tendency within 3 months before the first dose, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ or higher, or presence of vasculitis.
19. Active, known, or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, asthma requiring bronchodilators, etc.). Subjects in a stable state not requiring systemic immunosuppressive therapy are allowed.
20. Requirement for systemic treatment with corticosteroids (>10 mg/day prednisone equivalent) or other immunosuppressants within 14 days prior to study drug administration. Inhaled or topical steroids and adrenal replacement therapy at doses >10 mg/day prednisone equivalent are permitted in the absence of active autoimmune disease.
21. Prior treatment with other PD-1 antibodies or other immunotherapy targeting PD-1/PD-L1. Known history of severe allergy to any monoclonal antibody, anti-angiogenic targeted drugs, platinum agents, fluorouracil, or any component of the study drugs.
22. Requirement for long-term anticoagulation therapy with warfarin or heparin; requirement for long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).
23. Known history of psychotropic drug abuse or drug addiction. Pregnant or lactating women.
24. Any other factor considered by the investigator to be likely to lead to premature termination of the study, such as other severe diseases, significant laboratory abnormalities, or accompanying familial or social factors that may affect the subject's safety or the collection of trial data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | From the start of treatment until the date of first documented recurrence, metastasis, or death from any cause.ssessed regularly every 12 weeks (every 4 cycles) during treatment, then every 12 weeks until 24 months after treatment completion.
  The length of time after primary treatment for cancer ends that the patient survives without any signs or symptoms of that cancer. Tumor recurrence or metastasis will be determined based on radiological imaging (CT or MRI) and evaluated according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the start of treatment until the date of death from any cause, assessed every 3 months (±14 days) until 24 months after treatment completion.
  The length of time from the start of treatment that patients are still alive. It is a direct measure of the clinical benefit of the treatment.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 2 years
  The safety and tolerability of the combination therapy will be assessed by monitoring the type, frequency, severity, and relationship to study drugs of all adverse events and serious adverse events. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

OTHER OUTCOMES:
PD-L1 Expression Level in Tumor Tissue | Assessed at baseline (using archival tumor tissue obtained during prior surgical resection).
  An exploratory biomarker analysis to evaluate the level of programmed death-ligand 1 (PD-L1) protein expression in archival tumor tissue samples obtained during surgery and its potential association with clinical outcomes.